CLINICAL TRIAL: NCT04708509
Title: Extubation Advisor: Initial Implementation and Evaluation of a Novel Extubation Clinical Decision Support Tool
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2681
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Airway Extubation

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center interventional Phase 1 study to implement and evaluate perceptions of Extubation Advisor in consenting patients in the intensive care unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Wave form data from participants' spontaneous breathing trials (SBT) will be analyzed using Extubation Advisor (EA) to generate an EA report that provides clinical decision support regarding extubation.
  Interventions: Device: Extubation Advisor

INTERVENTIONS:
Device: Extubation Advisor — Participants undergoing a Spontaneous Breathing Trial (SBT) to assess readiness for extubation will be connected to a portable monitor displaying ECG, capnography, and other waveforms. This monitor will also be connected to a laptop containing the Extubation Advisor (EA) software. During the SBT, relevant patient information will be entered into the EA application and the EA application will record waveform data. When the SBT is complete, the EA application will analyze the waveform and patient data to generate a score summarizing the risk of extubation failure. A report will be generated and provided to the respiratory therapist and attending physician to help determine whether to proceed with extubation or not. Patients will be followed for 72 hours after extubation, when the clinical outcome case report form will be completed.

SUMMARY:
Expeditious, safe extubation is vitally important in the care of Intensive Care Unit (ICU) patients, as prolonged mechanical ventilation harms patients and failed extubation (i.e. re-intubation within 48 hrs) is associated with increased morbidity, mortality and costs. The urgent need to improve extubation failure is further highlighted by current observations suggesting that COVID-19 patients are at increased risk of both early and late extubation failure. The investigators previously found that decreased respiratory rate variability (indicative of reduced adaptability and/or increased stress) during Spontaneous Breathing Trials (SBTs) predicted extubation failure and outperformed the best available predictive indices. Combining this predictive analytic with standardized extubation readiness checklists and risk mitigation strategies, the investigators created the Extubation Advisor (EA). The investigators recently completed a single-center phase I mixed methods observational study (n=117) wherein there was demonstrated technical feasibility (i.e. ability to generate 92% EA of reports) and clinician acceptance of the EA tool. In the current open-label, multi-center interventional phase I study, the investigators will assess the feasibility and initial perceptions of EA implementation in the intensive care unit by (1) evaluating the feasibility of patient enrolment, data collection, and EA report generation, and (2) performing a mixed-methods analysis of critical care physician and respiratory therapist perceptions of EA. Findings from this study will inform a future randomized controlled trial assessing EA outcomes compared to standard of care, with the intent of aiding bedside decision-making, enhancing care delivery, and improving outcomes in critically ill patients with and without COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* In the Intensive Care Unit (ICU)
* Able to provide informed consent (through a surrogate)
* Invasive mechanical ventilation for > 48 hours
* Ready for spontaneous breathing test (SBT) for assessment for extubation
* At least partial reversal of the condition precipitating mechanical ventilation
* Stabilization of other organ systems
* Toleration of pressure support ventilation less than or equal to 14 cm H2O, (oxygen saturation (SpO2) greater than or equal to 90% with fraction of inspired oxygen (FiO2) less than or equal to 40% and positive end-expiry pressure (PEEP) less than or equal to 10cm H2O)
* Hemodynamic stability (low - phenylephrine less than 50 ug/min; norepinephrine less than 5 ug/min; dobutamine less than 5 ug/kg/min; milrinone less than 0.4 ug/kg/min - or no vasopressors)
* Stable neurological status (no deterioration in Glasgow coma score during prior 24 hours and, if measured, intracranial pressure (ICP) less than 20 mmHg)
* Intact airway reflexes (adequate cough with suctioning and a gag reflex)
* Normal sinus rhythm at the time of the SBT (no pacemaker)

Exclusion Criteria:

* Order not to re-intubate should the patient fail extubation
* Anticipated withdrawal of life support
* Known or suspected severe weakness (myopathy, neuropathy, or quadriplegia)
* Tracheostomy
* Prior extubation during current ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew JE Seely, MD, PhD, FRCSC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hryciw BN, Hudek N, Brehaut JC, Herry C, Scales N, Lee E, Sarti AJ, Burns KEA, Seely AJE. Extubation Advisor: Implementation and Evaluation of A Novel Extubation Clinical Decision Support Tool. J Intensive Care Med. 2025 Apr;40(4):418-426. doi: 10.1177/08850666241291524. Epub 2024 Oct 24. PMID 39444331

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Feasibility of Enrolling and Consenting Greater Than 50% of Eligible Patients
Description: Feasibility of patient enrolment and consent will be evaluated by determining if greater than 50% of eligible patients are enrolled and consented
Time Frame: Upon study completion, 4 months after study initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Evaluate Feasibility of Capturing Greater Than 75% of Wave Form Data
Description: Feasibility of wave form data capture will be evaluated by determining if greater than 75% of the time, wave form data is captured
Time Frame: Upon study completion, 4 months after study initiation
Measure: Number; unit: SBTs
Units Other Than Participants: SBTs
Arm/Group | Intervention Arm
Number analyzed (Participants) | 29
Number analyzed (SBTs) | 70
SBTs | 68

3. Primary Outcome: Evaluate Feasibility of Generating and Delivering Greater Than 80% of Extubation Advisor Reports to the Attending Physician
Description: Feasibility of Extubation Advisor report generation will be evaluated by determining if greater than 80% of the time, an extubation report is successfully generated and delivered to the attending physician
Time Frame: Upon study completion, 4 months after study initiation
Measure: Number; unit: EA reports delivered to attending MD
Units Other Than Participants: SBTs initiated
Arm/Group | Intervention Arm
Number analyzed (Participants) | 29
Number analyzed (SBTs initiated) | 70
EA reports delivered to attending MD | 55

ADVERSE EVENTS:
Time Frame: Adverse event (AE)/adverse device effect (ADE) data was collected from initiation of each spontaneous breathing trial (SBT) until 72 hours after exposure to the tool up to 28 days following enrolment.
Description: In this device study, for users or other persons, the definition of AE is restricted to events related to investigational medical devices, and considered as ADE. This definition includes AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational device, and includes any event resulting from use error or from intentional misuse of the investigational medical device.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT04708509/Prot_SAP_000.pdf